CLINICAL TRIAL: NCT02959983
Title: A Phase 4 Multicenter, Multinational, Prospective, Randomized, Placebo-Controlled, Double-Blinded Parallel Group Study to Assess Efficacy of Eluxadoline in the Treatment of Irritable Bowel Syndrome With Diarrhea (IBS-D) in Patients Who Report Inadequate Control of IBS-D Symptoms With Prior Loperamide Use (RELIEF)
Brief Title: Efficacy of Eluxadoline in the Treatment of Irritable Bowel Syndrome With Diarrhea in Patients With Inadequate Control of Symptoms With Prior Loperamide Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMO-US-GI-0429
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eluxadoline (Active Comparator): Eluxadoline 100 mg oral tablets twice daily (BID) with food for 12 weeks.
  Interventions: Drug: Eluxadoline
- Placebo (Placebo Comparator): Placebo matching eluxadoline oral tablets BID with food for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eluxadoline — Eluxadoline 100 mg oral tablets BID with food.
  Other Names: VIBERZI™
  Arms: Eluxadoline
Drug: Placebo — Placebo matching eluxadoline oral tablets BID with food.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of eluxadoline 100 milligrams (mg) twice a day (BID) versus placebo for the treatment of patients with Irritable Bowel Syndrome with Diarrhea (IBS-D) who report that the use of loperamide in the prior 12 months failed to provide control of their IBS-D symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of IBS-D, defined by the Rome III criteria as loose (mushy) or watery stools ≥25% and hard or lumpy stools ≤25% of bowel movements.
* Has had a colonoscopy performed within 5 years prior to Screening if they are at least 50 years of age, OR if they meet any of the following alarm features:

  1. Has documented weight loss within the past 6 months; or
  2. Has nocturnal symptoms; or
  3. Has a familial history of colon cancer; or
  4. Has blood mixed with their stool (excluding any blood from hemorrhoids)
* Patient reports use of loperamide in the 12 months prior to Screening for IBS-D symptoms and that loperamide did not provide adequate control of IBS-D symptoms.
* Has not used any loperamide rescue medication within 14 days prior to randomization.

Exclusion Criteria:

* Has a diagnosis of Irritable Bowel Syndrome (IBS) with a subtype of constipation IBS, mixed IBS, or unsubtyped IBS.
* Has a history of inflammatory or immune-mediated gastrointestinal (GI) disorders including inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis), microscopic colitis, or celiac disease.
* Has a history of diverticulitis within 3 months prior to screening.
* Has a documented history of lactose intolerance.
* Has a documented history of bile-acid malabsorption.
* Has a history of chronic or severe constipation or intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions.
* Has any of the following surgical history:

  1. Cholecystectomy or previously documented agenesis of gallbladder; or
  2. Any abdominal surgery within the 3 months prior to screening; or
  3. Major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post-surgery are allowed).
* Has a history of cholecystitis within 6 months before screening.
* Has a history of pancreatitis or structural diseases of the pancreas, including known or suspected pancreatic duct obstruction.
* Has a history of known or suspected biliary duct obstruction or sphincter of Oddi disease or dysfunction, excluding a history of gallstones.
* Has a history or current evidence of laxative abuse within 5 years prior to screening.
* Has documented evidence of cirrhosis.
* Has a history of cardiovascular events, including stroke, myocardial infarction, congestive heart failure, or transient ischemic attack within 6 months prior to screening.
* Has an unstable renal, hepatic, metabolic, or hematologic condition.
* Has a history of malignancy within 5 years before screening (except squamous and basal cell carcinomas and cervical carcinoma in situ).
* Has a history of human immunodeficiency virus infection.
* Has a history of Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision-defined substance dependency, excluding nicotine and caffeine, within 2 years prior to screening.
* Has a history of alcohol abuse, alcohol addiction, and alcoholism or drinks more than 3 alcoholic beverages per day.
* Has used aspirin or aspirin-containing medications (>325 mg of aspirin per day) or nonsteroidal anti-inflammatory drugs, when taken specifically for the symptoms of IBS, within 14 days of randomization.
* Has current (within 14 days of randomization) or expected use of any narcotic or opioid-containing agents, tramadol, docusate, enemas, GI preparations (including antacids containing aluminum or magnesium, antidiarrheal agents [except loperamide rescue medication after randomization]), antinausea agents, antispasmodic agents, bismuth, or prokinetic agents.
* Has current (within 28 days of randomization) use of rifaximin or other antibiotics (with the exception of topical antibiotics or a 1-day course with an antibiotic). Expected use of rifaximin or other antibiotics during the course of the study that is known at the time of randomization.
* Has an elective surgery planned or expects to need elective surgery at any time during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Jo, Study Director — Allergan
Locations (83):
- United States (76):
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - The Center for Clinical Trials, Saraland, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Med Investigations, Carmichael, California
  - GW Research Inc, Chula Vista, California
  - Diagnamics Inc, Encinitas, California
  - Behavioral Research Specialists, LLC, Irvine, California
  - Providence Clinical Research, North Hollywood, California
  - Shahram Jacobs MD INC., Sherman Oaks, California
  - Westlake Medical Research, Thousand Oaks, California
  - Upland Clinical Research, Upland, California
  - Advanced RX Clinicial Research Group, Inc., Westminster, California
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Digestive Care of N. Broward, Coral Springs, Florida
  - Homestead Medical Research, Homestead, Florida
  - Clinical Neuroscience Solutions Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Precision Clinical Research LLC, Lauderdale Lakes, Florida
  - Pharmax Research Clinic Inc., Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Ocean Blue Medical Research Center, Inc, Miami Springs, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Clinical Neuroscience Solutions Inc., Orlando, Florida
  - Clinical Research of West Florida Inc., Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - RNA America, LLC, Buford, Georgia
  - Northwestern University Feinbery School of Medicine, Chicago, Illinois
  - Pharmakon Inc, Evergreen Park, Illinois
  - Investigators Research, Brownsburg, Indiana
  - Radiant Research, Inc., Evansville, Indiana
  - Clinical Research Advantage Inc/Radiant Research Inc., Evansville, Indiana
  - Gtc Research, Shawnee Mission, Kansas
  - Investigative Clinical Research, Annapolis, Maryland
  - MGG Group Co. Inc. Chevy Chase Clinical Research, Chevy Chase, Maryland
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Clinical Research Insititute of Michigan LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Drug Trials Brooklyn, Brooklyn, New York
  - NY Scientific, Brooklyn, New York
  - Long Island Gastrointestinal Group LLP, Great Neck, New York
  - IMA Medical Research, PC, Kew Gardens, New York
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Peters Medical Research LLC, High Point, North Carolina
  - North State Clincial Research PLLC, Lenoir, North Carolina
  - Wake Research Associates LLC, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Buckeye Health and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Huber Heights, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - The Oregon Center for Clinical Investigations, INC., Salem, Oregon
  - Partners in Clinical Research, Cumberland, Rhode Island
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - CNS Healthcare, Memphis, Tennessee
  - Premier Family Physicians, Austin, Texas
  - Family Medicine Associate of Texas, Carrollton, Texas
  - Multi-Phase Trials LLC, San Antonio, Texas
  - Health Texas Research Institute, San Antonio, Texas
  - Discovery Clinical Trials - Stone Oak, San Antonio, Texas
  - Carl Meisner Medical Clinic, Sugar Land, Texas
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
- Canada (7):
  - Corunna Medical Research Centre, Corunna, Ontario
  - Manna Research, Etobicoke, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - University of Calgary, Calgary
  - Viable Clinical Research Corp., Nova Scotia
  - Centre de reserche St Louis, Québec
  - Dynamik Research Inc, Québec

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 660 participants were screened; 346 participants were randomized; 344 participants received at least 1 dose of study drug which comprises the safety population. Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study.
Period: Overall Study
Arm/Group | Eluxadoline | Placebo
Started | 172 | 174
Completed | 146 | 149
Not Completed | 26 | 25
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 12 | 9
Not completed — Other | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 7 | 12

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat population includes all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eluxadoline | Placebo | Total
Number analyzed (Participants) | 172 | 174 | 346
Age, Customized [Count of Participants; unit: Participants]
  <65 | 158 | 161 | 319
  ≥65 | 14 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 119 | 243
  Male | 48 | 55 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 41 | 74
  Not Hispanic or Latino | 139 | 133 | 272
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 144 | 141 | 285
  Black or African American | 20 | 26 | 46
  Asian | 7 | 3 | 10
  American Indian or Alaskan Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Composite Responders Based on Improvements From Baseline in Daily Worst Abdominal Pain And Daily Stool Consistency Scores
Description: Percentage of primary composite responders is defined as the percentage of participants who meet both of the following daily composite criteria for at least 50% of the days with diary entry: 1)Worst Abdominal Pain (WAP) score improved by ≥40% compared to Baseline. The participant records their WAP score in the past 24 hours each day in a daily patient diary where: 0=no pain to 10=worst imaginable pain. 2) Bristol Stool Score (BSS) <5; or the absence of a bowel movement if accompanied by ≥40% improvement in WAP compared to Baseline. The participant records their stool consistency each day in a daily patient diary using the BSS on a scale from 1 (hard stool) to 7 (watery stool).
Time Frame: Baseline, Weeks 1 to 12
Population: The Intent-to-Treat population includes all randomized patients.
Measure: Number; unit: percentage of participants
Arm/Group | Eluxadoline | Placebo
Number analyzed (Participants) | 172 | 174
percentage of participants | 22.7 | 10.3
Statistical Analysis 1: Comparison: Eluxadoline vs Placebo; Overall Weeks 1-12; Test type: Superiority; p = 0.0022, Chi-squared

2. Secondary Outcome: Percentage of Stool Consistency Responders
Description: Percentage of stool consistency responders is defined as the percentage of participants who meet the daily stool consistency response criteria: BSS <5; or the absence of a bowel movement if accompanied by ≥40% improvement in WAP compared to Baseline for ≥50% of days with daily patient diary entries over a certain time period. The participant records their stool consistency each day in a daily patient diary using the BSS on a scale from 1 (hard stool) to 7 (watery stool). A participant must have had a minimum of 20 days of diary entries over any 4-week interval.
Time Frame: Weeks 1 to 12 and 4-week intervals (Weeks 1 to 4, Weeks 5 to 8 and Weeks 9 to 12)
Population: The Intent-to-Treat population includes all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Eluxadoline | Placebo
Number analyzed (Participants) | 172 | 174
Percentage of Participants
  Overall Weeks 1 to 12 | 27.9 | 16.7
  Weeks 1 to 4 | 24.4 | 12.6
  Weeks 5 to 8 | 30.8 | 20.1
  Weeks 9 to 12 | 29.7 | 25.3
Statistical Analysis 1: Comparison: Eluxadoline vs Placebo; Overall Weeks 1 to 12; Test type: Superiority; p = 0.0119, Chi-squared
Statistical Analysis 2: Comparison: Eluxadoline vs Placebo; Weeks 1 to 4; Test type: Superiority; p = 0.0048, Chi-squared
Statistical Analysis 3: Comparison: Eluxadoline vs Placebo; Weeks 5 to 8; Test type: Superiority; p = 0.0207, Chi-squared
Statistical Analysis 4: Comparison: Eluxadoline vs Placebo; Weeks 9 to 12; Test type: Superiority; p = 0.3700, Chi-squared

3. Secondary Outcome: Percentage of Pain Responders
Description: Percentage of pain responders is defined as the percentage of participants who meet the daily pain response criteria: WAP score improved by ≥40% compared to Baseline for ≥50% of days with diary entries over a certain time period. The participant records their WAP score in the past 24 hours each day in a daily diary where: 0=no pain to 10=worst imaginable pain. A participant must have had a minimum of 20 days of diary entries over any 4-week interval.
Time Frame: Baseline, Weeks 1 to 12 and 4-week intervals (Weeks 1 to 4, Weeks 5 to 8 and Weeks 9 to 12)
Population: The Intent-to-Treat population includes all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Eluxadoline | Placebo
Number analyzed (Participants) | 172 | 174
Percentage of Participants
  Overall Weeks 1 to 12 | 43.6 | 31.0
  Weeks 1 to 4 | 30.2 | 25.9
  Weeks 5 to 8 | 45.9 | 31.6
  Weeks 9 to 12 | 44.8 | 35.1
Statistical Analysis 1: Comparison: Eluxadoline vs Placebo; Overall Weeks 1 to 12; Test type: Superiority; p = 0.0174, Chi-squared
Statistical Analysis 2: Comparison: Eluxadoline vs Placebo; Weeks 1 to 4; Test type: Superiority; p = 0.3832, Chi-squared
Statistical Analysis 3: Comparison: Eluxadoline vs Placebo; Weeks 5 to 8; Test type: Superiority; p = 0.0052, Chi-squared
Statistical Analysis 4: Comparison: Eluxadoline vs Placebo; Weeks 9 to 12; Test type: Superiority; p = 0.0619, Chi-squared

4. Secondary Outcome: Percentage of Monthly Composite Responders
Description: Percentage of monthly composite responders is defined as the percentage of participants who meet the daily composite response criteria for at least 50% of days with diary entry for a minimum of 20 days during each 4-week interval (weeks 1 to 4, 5 to 8, and 9 to 12). Composite response includes both of the following criteria: 1) WAP score improved by ≥40% compared to Baseline. The participant records their WAP score in the past 24 hours each day in a daily patient diary where: 0=no pain to 10=worst imaginable pain. 2) BSS <5; or the absence of a bowel movement if accompanied by ≥40% improvement in WAP compared to Baseline. The participant records their stool consistency each day in a daily patient diary using the BSS on a scale from 1 (hard stool) to 7 (watery stool).
Time Frame: Weeks 1 to 4, 5 to 8, and 9 to 12
Population: The Intent-to-Treat population includes all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Eluxadoline | Placebo
Number analyzed (Participants) | 172 | 174
Percentage of Participants
  Weeks 1-4 | 14 | 6.9
  Weeks 5-8 | 26.7 | 14.9
  Weeks 9-12 | 30.8 | 16.7
Statistical Analysis 1: Comparison: Eluxadoline vs Placebo; Weeks 1-4; Test type: Superiority; p = 0.0330, Chi-squared
Statistical Analysis 2: Comparison: Eluxadoline vs Placebo; Weeks 5 to 8; Test type: Superiority; p = 0.0063, Chi-squared
Statistical Analysis 3: Comparison: Eluxadoline vs Placebo; Weeks 9 to 12; Test type: Superiority; p = 0.0018, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The Safety Population will include all patients enrolled who received at least 1 dose of study drug. Safety data will be analyzed using the safety population.
Arm/Group | Eluxadoline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/173
Serious Adverse Events (participants affected / at risk) | 1/171 | 3/173
Other Adverse Events (participants affected / at risk) | 10/171 | 5/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline (N=171) | Placebo (N=173)
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eluxadoline (N=171) | Placebo (N=173)
Nausea (Gastrointestinal disorders) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT02959983/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT02959983/SAP_001.pdf